CLINICAL TRIAL: NCT07049796
Title: Impact of a Pharmaceutical Interview on the Initiation of Opioid Treatment for Acute Non-cancer Pain in Short Stay Hospitalization Units (UHCD) and Downstream Hospitalization Units (UHA) of Adult Emergency Departments
Brief Title: Impact of a Pharmaceutical Interview at the Initiation of Opioid Treatment for Acute Non-cancer Pain
Acronym: OPI-HOME
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/152/OB; N° IDRCB : 2021-A01246-35 (Other: ANSM)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-01

CONDITIONS: Interviews
Keywords: Impact and feasibility of a pharmaceutical interview; opioid treatment
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort including patients with opioid analgesic treatment upon discharge from hospital

SUMMARY:
In adult emergency departments, the number of admissions for adverse effects related to opioid use is constantly increasing. However, the massive flow of patients, lack of time, and rapid rotation of physicians in this department do not favor the transmission of in-depth information on the proper use of these therapies to the patient. In addition, this therapeutic class tends to worry patients. Public authorities as well as the medical profession are concerned about the potential adverse effects of morphine, but also the potential misuse, or even overdose, which can be fatal for the patient. Interventions by the community pharmacist in the fight against this misuse seem interesting, but an intervention upstream of potential problems of proper use seems even more relevant to us. Recent studies have shown the strong interest of the pharmacist in a multidisciplinary team on pain and opioids, both at the local level with studies conducted at the Rouen University Hospital by C. LATTARD et al. in rheumatology and E.BARAT et al. in outpatient surgery. It also appears that knowledge on the subject is satisfactory. Work conducted by Winstanley et al. shows that the intervention of a pharmacist in the emergency department seems relevant in terms of patient knowledge and satisfaction, and entirely feasible.

DETAILED DESCRIPTION:
This study aims to measure the clinical impact of a hospital pharmacist when initiating opioid treatment for acute non-cancer pain in the Short Stay Hospitalization Units (UHCD) and Downstream Hospitalization Units (UHA) of the adult emergency department at Rouen University Hospital.

Pharmacy interviews will be offered to patients meeting the inclusion criteria. These 15- to 30-minute interviews will aim to present the tools implemented by the Rouen University Hospital pharmacy team. Several topics will be discussed, including: treatment optimization, potential adverse effects and what to do if they occur, the differences between immediate-release (IR) and extended-release (LP) forms, what to do if a dose is missed, the risks of overdose and addiction, and storage methods.

The objective of this project is, firstly, to improve patient satisfaction with their care and, secondly, to better understand the treatment, thus enabling more optimal use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years old)
* Patient admitted to the following departments: Downstream Hospitalization Unit (UHA) and Short-Term Hospitalization Unit (UHCD)
* Independent patient or assisted by close family (who can receive information with the patient)
* Initiation of opioid treatment for acute non-cancer pain during their stay in the Emergency Department, UHA, or UHCD or shortly before (<7 days)
* Patient speaks French
* Presence of the clinical pharmacist in the relevant departments

Exclusion Criteria:

* Patient with drug addiction
* Patient under guardianship/guardianship
* Patient transferred to rheumatology
* Patient already on opioid treatment for ≥ 7 days
* Patient refuses
* Patient assisted by a nurse at home or a caregiver not present during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients over 18 years of age with opioid analgesic treatment upon discharge from hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of satisfaction with a pharmaceutical interview for acute pain | Day 7
  To assess satisfaction with pharmaceutical care for acute non-cancer pain in short-term hospitalization units (UHCD) and emergency downstream hospitalization units (UHA) during a telephone call to the patient 7 days after discharge from hospital. This satisfaction will be quantified as a percentage from 0 to 100%.

SECONDARY OUTCOMES:
Evaluation of the relevance and effectiveness of pharmaceutical maintenance against pain | Day 3
  Patient satisfaction with pharmaceutical pain management on day 3 will be assessed during a telephone call to the patient 3 days after discharge from hospital. This satisfaction will be quantified as a percentage from 0 to 100%.
Evaluation of the relevance and effectiveness of pharmaceutical maintenance against pain | Day 3 and Day 7
  The average pain assessment on admission, discharge, day 3 and day 7 will be evaluated using a numerical scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna JR RAYMOND, Doctor, Study Director — University Rouen Hospital
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.